CLINICAL TRIAL: NCT03873779
Title: A Feasibility Study to Explore the Safety and Efficacy of Cryolipolysis Followed by Radiofrequency Treatment for Submental and Submandibular Contouring
Brief Title: CoolSculpting and RF for the Submental
Acronym: CRT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zeltiq Aesthetics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ZA18-002
Record Dates: First submitted 2018-12-18; First posted 2019-03-13 (Actual); Results first posted 2025-03-10 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-02

CONDITIONS: Body Fat Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Cryolipolysis Followed by Radiofrequency Treatment (Experimental)
  Interventions: Device: The ZELTIQ System

INTERVENTIONS:
Device: The ZELTIQ System — Participants received cryolipolysis treatment in submental and submandibular areas using the CoolSculpting System and CoolMini applicator for fat layer reduction on Day 0, which was followed with a radiofrequency treatment performed 12 weeks after CoolSculpting.

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of sequential use of CoolSculpting (Cryolipolysis) and radiofrequency treatment of the submental and submandibular area.

ELIGIBILITY:
Inclusion Criteria

* Male or female subjects ≥22 years of age and ≤65 years of age.
* Treatment area skin fold thickness > 1cm (measured by caliper).
* Dissatisfaction with the treatment area expressed by the subject as a rating of 0, 1 or 2 using the Subject Self Rating Scale (SSRS) as determined at Screening visit.
* No weight change exceeding 5% of body weight in the preceding month.
* Agreement to maintain his/her weight (i.e., within 5%) by not making any major changes in diet or exercise routine during the course of the study.
* Subject has signed a written informed consent form

Exclusion Criteria

* Body Mass Index ≥ 46.2 as determined at screening.
* Excessive skin laxity in the treatment area for which reduction of subcutaneous fat may, in the opinion of the investigator, result in an unacceptable aesthetic result.
* Prominent platysmal bands at rest which may interfere with assessment of treatment area.
* Evidence of any cause of enlargement in the treatment area other than localized subcutaneous fat, such as swollen lymph nodes or ptotic submandibular glands.
* Significant enlargement on the anterior neck that may prevent the proper placement of the applicator e.g. enlarged thyroid glands.
* Treatment with dermal fillers, chemical peels, radiofrequency or laser procedures that may affect contour in the treatment area within the past 6 months.
* Botulinum toxin, deoxycholic acid, or other aesthetic drug injections within the treatment area in the past 6 months.
* History of facial nerve paresis or paralysis (such as Bell's palsy).
* History of a fat reduction procedure (e.g., liposuction, surgery, lipolytic agents, etc.) or implant in or adjacent to the area of intended treatment.
* History of prior neck surgery, or prior surgery in the area of intended treatment.
* Current infection in and adjacent to treatment area.
* Known history of cryoglobulinemia, cold urticaria, cold agglutinin disease or paroxysmal cold hemoglobinuria.
* Known history of Raynaud's disease, or any known condition with a response to cold exposure that limits blood flow to the skin.
* History of bleeding disorder or is taking any medication that in the investigator's opinion may increase the subject's risk of bruising.
* Currently taking or has taken diet pills or weight control supplements within the past month.
* Any dermatological conditions, such as scars in the location of the treatment area that may interfere with the treatment or evaluation.
* Active implanted device such as a pacemaker, automatic implantable cardioverter/defibrillator (AICD), drug delivery system, or any other implantable electrical device.
* Pregnant or intending to become pregnant in the next 6 months.
* Lactating or has been lactating in the past 6 months.
* Unable or unwilling to comply with the study requirements including remaining clean shaven for all study visits.
* Currently enrolled in a clinical study of an unapproved investigational drug or device.
* Any other condition or laboratory value that would, in the professional opinion of the investigator, potentially affect the subject's response or the integrity of the data or would pose an unacceptable risk to the subject.

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2018-12-18 (Actual); Primary Completion 2019-06-18 (Actual); Study Completion 2019-06-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Innovation Research Center, Pleasanton, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A separate cohort was initially planned for radiofrequency treatment immediately following cryolipolysis at the same visit, however no participants were enrolled in this cohort.
Groups:
- Cryolipolysis Followed by Radiofrequency Treatment: Participants received cryolipolysis treatment in submental and submandibular areas using the CoolSculpting System and CoolMini applicator for fat layer reduction on Day 0, which was followed with a radiofrequency treatment performed 12 weeks after CoolSculpting.
Period: Overall Study
Arm/Group | Cryolipolysis Followed by Radiofrequency Treatment
Started | 8
Received Cryolipolysis Treatment | 8
Received Radiofrequency Treatment | 7
Completed | 7
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: The Safety Population consisted of all participants who received at least one study treatment.
Arm/Group | Cryolipolysis Followed by Radiofrequency Treatment
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Black or African American | 0
  Native Hawaiian or Other Pacific Islander | 0
  White | 3
  Other | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Unanticipated Adverse Device Effects (UADEs)
Description: UADEs were defined as any serious adverse effect on health and safety or any life-threatening problem or death caused by, or associated with a device, if that effect, problem, or death was not previously identified in nature, severity, or degree of incidence in the investigational plan or application, or any other unanticipated serious problem associated with a device that relates to the rights, safety, or welfare of participants.
Time Frame: From date of first treatment to 12 weeks after final treatment (up to 24 weeks)
Population: The Safety Population consisted of all participants who received at least one study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Cryolipolysis Followed by Radiofrequency Treatment
Number analyzed (Participants) | 8
Participants | 0

2. Primary Outcome: Number of Participants With Global Aesthetic Improvement Per Independent Physician Review of Photographs Based on Investigator Global Aesthetic Improvement Scale (GAIS-Independent)
Description: Photos obtained during the study were reviewed by an independent physician reviewer who entered assessments according to the Global Aesthetic Improvement Scale (GAIS). The GAIS had outcome choices of "very much improved", "much improved", "improved", "no change", "worse", "much worse", or "very much worse", with "very much improved" representing the most aesthetic improvement. Reported here is the sum of participants who were assessed as improved ("Very Much Improved," "Much Improved", and "Improved").
Time Frame: Baseline, 12 weeks post radiofrequency treatment
Population: The Per-protocol population (PP) consisted of all participants who received both CoolSculpting and radiofrequency treatment, and had a weight change of no more than 5 percent at the time of the 12-week post final treatment visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Cryolipolysis Followed by Radiofrequency Treatment
Number analyzed (Participants) | 6
Participants | 2

3. Secondary Outcome: Percent Change From Baseline in Fat Layer Thickness
Description: Fat layer thickness was measured using a caliper at the center of the treatment area.
Time Frame: Baseline, 12 weeks post radiofrequency treatment
Population: The PP population consisted of all participants who received both CoolSculpting and radiofrequency treatment, and had a weight change of no more than 5 percent at the time of the 12-week post final treatment visit.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Cryolipolysis Followed by Radiofrequency Treatment
Number analyzed (Participants) | 6
percent change | -31.9 (9.4)

4. Secondary Outcome: Number of Participants With Improvement Based on Subject-graded Global Aesthetic Improvement Scale (SGAIS)
Description: Participants rated improvement in their treatment areas based on the SGAIS. The SGAIS had outcome choices of "very much improved", "much improved", "improved", "no change", "worse", "much worse", or "very much worse", with "very much improved" representing the most aesthetic improvement. Reported here is the sum of participants who reported as improved ("Very Much Improved," "Much Improved", and "Improved").
Time Frame: Baseline, 12 weeks post radiofrequency treatment
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Cryolipolysis Followed by Radiofrequency Treatment
Number analyzed (Participants) | 6
Participants | 6

5. Secondary Outcome: Number of Participants With Positive Response in Subject Self-Rating Scale (SSRS) Score
Description: Participants assessed their own satisfaction with their face and chin using the SSRS. The SSRS is a participants self-rating scale, scored on a 7-point scale with 0=extremely dissatisfied, 1=dissatisfied, 2=slightly dissatisfied, 3=neither satisfied nor dissatisfied, 4=slightly satisfied, 5=satisfied, and 6=extremely satisfied, with 6 representing higher participant satisfaction. Reported here is the number of participants with a score of 4 or higher, indicating satisfaction.
Time Frame: Baseline, 12 weeks post radiofrequency treatment
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Cryolipolysis Followed by Radiofrequency Treatment
Number analyzed (Participants) | 6
Participants | 5

6. Secondary Outcome: Number of Participants With Positive Response on Subject Satisfaction Questionnaire
Description: Participants reported their satisfaction with aspects of treatment on a written questionnaire which included a 5-point Likert scale ranging from -2 to 2, with -2 representing more negative response and 2 representing more positive response. Reported here are the numbers of participants with responses of 1 or 2, indicating a positive response, to the following categories: Comfort of Treatment Procedure, How Visible is Fat Reduction, Overall Effect from the Procedure, Overall Satisfaction with Treatment from the Procedure to the Result, Made Me Look More Youthful, Made My Chin Look More Toned, Feel Less Self-Conscious About Chin Fat, Overall Appearance Has Improved.
Time Frame: Baseline, 12 Weeks Post Radiofrequency Treatment
Population: The Per-protocol population consisted of all participants who received at least 1 study treatment and had a weight change of no more than 5 percent at the time of the 12-week post final treatment visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Cryolipolysis Followed by Radiofrequency Treatment
Number analyzed (Participants) | 6
Participants
  Comfort of Treatment Procedure | 3
  How Visible is Fat Reduction | 4
  Overall Effect from the Procedure | 3
  Overall Satisfaction with Treatment, from the Procedure to the Result | 5
  Made Me Look More Youthful | 4
  Made My Chin Look More Toned | 4
  Feel Less Self-Conscious About Chin Fat | 4
  Overall Appearance Has Improved | 4

ADVERSE EVENTS:
Time Frame: From date of first treatment to 12 weeks after final treatment (up to 24 weeks)
Description: The Safety Population consisted of all participants who received at least one study treatment.
Arm/Group | Cryolipolysis Followed by Radiofrequency Treatment
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-19): https://cdn.clinicaltrials.gov/large-docs/79/NCT03873779/Prot_SAP_000.pdf